CLINICAL TRIAL: NCT05809869
Title: A Phase 2 Study on Immune Checkpoint Inhibitors and Radioembolisation for Previously Untreated Metastatic Hepatocellular Carcinoma
Brief Title: Immunotherapy and Radioembolisation for Metastatic Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 22-729
Record Dates: First submitted 2023-02-26; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Immune checkpoint inhibitors and radioembolisation for previously untreated metastatic hepatocellular carcinoma
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab in combination with tremelimumab and radioembolisation (Experimental): 1. Tremelimumab 300 mg intravenous infusion on week 1 only
  2. Durvalumab 1500mg intravenous infusion on week 1, 5, 9, 13, 17, 21 and 25, for a total of 7 cycles
  3. Radioembolisation with yttrium-90 microspheres on week 2 only
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Radiation: Yttrium-90 radioembolisation

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg intravenous infusion on week 1, 5, 9, 13, 17, 21 and 25 for a total of 7 cycles
  Other Names: MEDI4736
Drug: Tremelimumab — Tremelimumab 300mg intravenous infusion on week 1 only.
  Other Names: Imjudo
Radiation: Yttrium-90 radioembolisation — Yttrium-90 radioembolisation on week 2 only.

SUMMARY:
Hepatocellular carcinoma is one of the most intractable primary malignancies in the hepatobiliary and pancreatic tract with a poor overall survival worldwide. Unfortunately, the vast majority of hepatocellular carcinoma patients suffer from advanced unresectable or metastatic disease at diagnosis. Currently targeted therapy alone, or in combination with anti-vascular endothelial growth factor antagonist, is the standard first-line treatment for metastatic hepatocellular carcinoma.

On the other hand, there is growing evidence suggesting that radiation therapy (external or internal) with or without immune checkpoint inhibitors can produce or even augment abscopal effect in which the tumours away from the radiation field also show significant tumour shrinkage. The underlying mechanism of eliciting abscopal effect includes the increased antigen presentation by the myeloid cells within the tumour stroma leading to enhanced tumour cell killing. Previous case reports showed that radiation therapy alone can induce abscopal effect in mice and human models. However, a robust and concrete evidence of abscopal effect with combinational immune checkpoint inhibitors and radioembolisation or external radiation therapy in hepatocellular carcinoma is still lacking.

This study investigates the efficacy and safety of immune checkpoint inhibitors and radioembolisation as first-line treatment for previously untreated metastatic hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is one of the most intractable primary malignancies in the hepatobiliary and pancreatic tract with a poor overall survival worldwide. Surgery in the form of hepatectomy or liver transplantation provides the best chance of cure for early-stage disease. Unfortunately, the vast majority of hepatocellular carcinoma patients suffer from advanced unresectable or metastatic disease at diagnosis. Currently targeted therapy alone, or in combination with anti-vascular endothelial growth factor antagonist, is the standard first-line treatment for metastatic hepatocellular carcinoma.

On the other hand, there is growing evidence suggesting that radiation therapy (external or internal) with or without immune checkpoint inhibitors can produce or even augment abscopal effect in which the tumours away from the radiation field also show significant tumour shrinkage. The underlying mechanism of eliciting abscopal effect includes the increased antigen presentation by the myeloid cells within the tumour stroma leading to enhanced tumour cell killing. Previous case reports showed that radiation therapy alone can induce abscopal effect in mice and human models. However, a robust and concrete evidence of abscopal effect with combinational immune checkpoint inhibitors and radioembolisation or external radiation therapy in hepatocellular carcinoma is still lacking.

This phase 2 single-arm study will investigate the efficacy and safety of combination of immune checkpoint inhibitors and radioembolisation for previously untreated metastatic hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic hepatocellular carcinoma (HCC) confirmed by radiological findings with contrast-enhanced triphasic CT scan of the liver and/or MRI scan of the abdomen, without or without histological/cytological confirmation or elevation of serum alpha-feto protein.
* Must be of age 18 years or above.
* Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at study entry.
* Must be eligible to receive immune checkpoint inhibitor and yttrium-90 microsphere injection.
* Must have baseline efficacy images with CT or MRI and measurable target lesions in the liver according to RECIST 1.1 and mRECIST, taken within 28 days prior to the start of immune checkpoint inhibitor.
* Must be able to provide written informed consent.
* Adequate serum hematological functions defined as:

Absolute neutrophil count (ANC) ≥1.0 x 10^9/l Platelet ≥75 x 10^9/l Haemoglobin ≥9 g/dL

* Adequate serum biochemistry functions defined as:

Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>> Serum aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤2.5 times of institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5 times of ULN

Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment or 5 half-lives, whichever is shorter.
* Has a diagnosis of severe active scleroderma, lupus, other rheumatologic or autoimmune disease within the past 3 months before study recruitment. Patients with a documented history of clinically severe autoimmune disease or a syndrome requiring systemic steroids or immunosuppressive agents will not be allowed on this study. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement are not excluded from this study.
* Has had a prior monoclonal antibody, immunotherapy or immune checkpoint inhibitors before recruitment into this study.
* Has had prior chemotherapy or targeted small molecule therapy (including sorafenib or other anti-vascular endothelial growth factor inhibitor) within 3 weeks prior to administration of the study drug or who has not recovered (i.e., grade ≤1 or at baseline) from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, indolent lymphomas, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known carcinomatous meningitis (also known as leptomeningeal carcinomatosis).
* Has an active infection requiring intravenous systemic therapy or hospital admission.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality, including psychiatric or substance abuse disorder, that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 31 weeks after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Routine checking for Anti-HIV1 or Anti-HIV2 is not mandatory.
* Untreated hepatitis B infection. Patients with chronic hepatitis B infection (defined as HBsAg positive) are eligible if they have started anti-viral therapy for at least 1 month and is continuing anti-viral treatment throughout the whole duration of this study.
* Has experienced Grade 4 toxicity on treatment with prior radiation.
* Has experienced grade 3-4 intracranial toxicity (hypophysitis or central nervous system toxicity) with either prior intracranial radiation, anti-programmed cell death-1 (PD-1), or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor therapy.
* Is taking >4mg/day of dexamethasone or its equivalent at the start of immunotherapy or has required >4mg/day of dexamethasone or its equivalent for 3 consecutive days within 1 week of starting treatment.
* Allergies and adverse drug reaction to the following: History of allergy to study drug components; History of severe hypersensitivity reaction to any monoclonal antibody.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study medication. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

(A) Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) (B) Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent (C) Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Best objective response | 3 years
  Best objective response
Rate of abscopal effect | 3 years
  Rate of abscopal effect, which is defined as the rate of objective response of tumour sites outside the liver after radioembolisation and immune checkpoint inhibitor therapy

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival
Overall survival | 3 years
  Overall survival
Incidence of treatment-related side effects | 3 years
  Incidence of treatment-related side effects as determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Local control rate | 3 years
  Local control rate, which is defined as the percentage of tumour sites in the liver without evidence of progressive disease after radioembolisation and immune checkpoint inhibitor therapy
Distant control rate | 3 years
  Distant control rate, which is defined as the percentage of tumour sites outside the liver without evidence of progressive disease after radioembolisation and immune checkpoint inhibitor therapy

CONTACTS AND LOCATIONS:
Overall Officials: Victor Ho-Fun Lee, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.